CLINICAL TRIAL: NCT00350805
Title: Relating the 'Experienced Present' With the Mechanisms of Neuronal Function: A Comparative Study in Patients With Schizophrenia and Healthy Controls Using Psychophysical and Neurophysiological Methods
Brief Title: Measuring Time Windows in Patients With Schizophrenia and Healthy Controls
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other); Institut de Physique Biologique de Strasbourg (Unknown)
Responsible Party: Sponsor
Other Study IDs: 3494
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Time perception; Cortical synchronization; Electroencephalography
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy volunteers
  Interventions: Procedure: EEG
- Patients
  Interventions: Procedure: EEG

INTERVENTIONS:
Procedure: EEG — One 20 minutes session

SUMMARY:
Abnormalities in the ability to distinguish events in time may have a great impact on everyday life. The main objective of the study is to evaluate the magnitude of the temporal windows in schizophrenia, i.e. the time interval during which two events are perceived as synchronous. The investigators test the hypothesis that these temporal windows are enlarged, and check the relationship between this impairment and disorganization symptoms, in order to explore the link between this cognitive impairment and clinical symptoms. They explore also the neurobiological bases of the impairment by means of electroencephalogram (EEG) recordings. Event-related potentials (N50) will reveal whether or not the coding of the stimuli has the same temporal characteristics in patients and controls. The distribution and amplitude of oscillatory activities will be analyzed as a function of the synchronous or asynchronous response of the subject, thus allowing to explore the links between synchrony perception and neuronal synchronization phenomena.

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia (DSM-IV criteria)
* Healthy controls matched with patients on age, sex and education level
* Age between 18 and 50
* Informed consent signed
* No severe somatic illness
* No invalidating sensory disease
* No drug abuse, as defined by DSM-IV criteria
* No general anesthesia in the past 3 months
* No intake of drug affecting the CNS, except for patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Primary care clinic, residents of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne GIERSCH, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (3):
- France (3):
  - Service de Psychiatrie Adulte & INSERM U841, Hôpital Albert Chenevier et Henri Mondor (AP-HP), Créteil
  - Centre Hospitalier de Rouffach, Rouffach
  - INSERM U666 - Département de Psychiatrie - Hôpitaux Universitaires de Strasbourg, Strasbourg